CLINICAL TRIAL: NCT05041400
Title: Distribution of Knee Isokinetic Angle-specific Moments and Ratios: Searching for Normative Values in Healthy Subjects
Brief Title: Distribution of Knee Isokinetic Angle-specific Moments and Ratios
Acronym: MOMANGLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/21/0251
Record Dates: First submitted 2021-09-02; First posted 2021-09-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Musculoskeletal Diseases
Keywords: knee isokinetic angle
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy subjects (Other): Evaluation carried out on a BIODEX S4 Pro isokinetic dynamometer after a standardised 10-minute warm-up on this same dynamometer .
  The measurement range will be from 0° (full extension) to 90° of flexion for each knee, providing 91 degrees of measurement.
  Interventions: Other: Evaluation of the strength of knee flexors and extensors

INTERVENTIONS:
Other: Evaluation of the strength of knee flexors and extensors — Each participant will benefit from a clinical evaluation and an evaluation of the strength of knee flexors and extensors using an isokinetic dynamometer after a 10-minute warm up.

SUMMARY:
The quantification of the strength-producing capacity of the knee joint muscles by isokinetic measurement is one of the most widely used tools for monitoring and deciding whether to return to sport after ACL reconstruction. However, the isokinetic evaluation performed in current practice does not exploit all the measures offered by this exploration technique, which can lead to errors in analysis and interpretation of the results and underestimate its ability to predict a return to sport under optimal conditions. Recently, more complete analysis models than those currently in use and integrating the moment-angle relationship have thus proposed the use of functional ratios sweeping the whole amplitude of the knee joint. Baumgart proposed an analysis of the variation of isokinetic force moments at each angle after ligamentoplasty. This approach seems to be the future of isokinetic performance analyses, but for the moment this has only been used in pathological populations and on small numbers of patients (less than 40). There are therefore no reference values in healthy subjects.

DETAILED DESCRIPTION:
Rupture of the anterior cruciate ligament is a common sports trauma injury, frequently leading to a surgical intervention. However, despite the extensive scientific literature on the subject, return to sports at a lower level is common, sometimes to the point of giving up pivoting sports. Current rehabilitation strategies and the means used tend to limit their effectiveness, as do the batteries of tests for returning to sport .

One of the most widely used assessments for monitoring and decision-making on return to sport after ACL reconstruction is the quantification of the strength production capacity of the knee joint muscles by isokinetic measurement. However, the isokinetic evaluation carried out in current practice does not exploit all the measures offered by this exploration technique, which can lead to errors in the analysis and interpretation of the results . This discrepancy between the possibilities offered by this tool and its current exploitation may underestimate its capacity to predict a return to sport under optimal conditions .

In clinical practice, the analysis is reduced to the consideration of two indices: the peak torques of the extensor and flexor muscles of the knee, which are compared between the two legs (right and left sides), and the ratio between the torque peak of the flexor muscles and that of the extensor muscles, this ratio being considered as a control of joint balance. More comprehensive analysis models than those currently in use and integrating the moment-angle relationship have thus proposed the use of functional ratios sweeping the knee's joint range of motion. Baumgart has proposed an analysis of the variation of isokinetic force moments at each angle after ligamentoplasty . This approach seems to be the future of isokinetic performance analyses, but has so far only been used in pathological populations and on small numbers of patients (less than 40). There are therefore no reference values in healthy subjects. The search for reference values for the torque of the muscles of the knee over the entire angular range of motion represents an important line of research to improve the objective evaluation of the neuromuscular performance of the knee and the return to sport of patients, particularly following ACL reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects,
* Practicing a regular activity with a minimal activity of two trainings and one competition per week,
* Practicing this activity from at least 8 continuous weeks,
* Affiliated or benefiting from public health services.

Exclusion Criteria:

* Person presenting any of these conditions: professional player / athlete,
* patient with systemic pathology or treatment affecting the musculoskeletal system, patient with a history of traumatic pathology or any pathology requiring orthopaedic/surgical treatment of the knee and/or hip and/or spine,
* patient having a contraindication to an isokinetic test (disabling pain, progressive pathological process, unconsolidated fracture, unbalanced cardiovascular pathology), protected patient (adults under guardianship or other legal protection, deprived of their liberty by judicial or administrative decision), Pregnant and/or breastfeeding women.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Distribution of knee isokinetic angle | 1 DAY
  The primary outcome will be composed of the following elements:(1)- a curve representing the distribution of the mean (and confidence interval) of the normative values of the knee flexors/extensors ratio at each angle on the tested amplitude, (2) a curve representing the distribution of the mean (and confidence interval) of the normative values of the right/left ratio at each angle on the tested amplitude,(3) a curve representing the distribution of the mean (and confidence interval) of the normative values of peak torque (normalized by subject mass) produced by the flexors and extensors at each angle over the amplitude tested, (4)- the distribution of the mean (and confidence interval) of the right/left differential on the value of the peak torque on the flexors and extensors and its angle of occurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Marc-Antoine DEMARET, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Marc Antoine DEMARET, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ardern CL, Taylor NF, Feller JA, Webster KE. Fifty-five per cent return to competitive sport following anterior cruciate ligament reconstruction surgery: an updated systematic review and meta-analysis including aspects of physical functioning and contextual factors. Br J Sports Med. 2014 Nov;48(21):1543-52. doi: 10.1136/bjsports-2013-093398. Epub 2014 Aug 25. PMID 25157180
- [Background] Gokeler A, Welling W, Zaffagnini S, Seil R, Padua D. Development of a test battery to enhance safe return to sports after anterior cruciate ligament reconstruction. Knee Surg Sports Traumatol Arthrosc. 2017 Jan;25(1):192-199. doi: 10.1007/s00167-016-4246-3. Epub 2016 Jul 16. PMID 27423208
- [Background] Baumgart C, Welling W, Hoppe MW, Freiwald J, Gokeler A. Angle-specific analysis of isokinetic quadriceps and hamstring torques and ratios in patients after ACL-reconstruction. BMC Sports Sci Med Rehabil. 2018 Dec 6;10:23. doi: 10.1186/s13102-018-0112-6. eCollection 2018. PMID 30534382